CLINICAL TRIAL: NCT00591019
Title: Use of Modafinil in the Treatment of Tinnitus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early due to lack of change in primary and secondary outcome measures.
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: # 65171
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-09

CONDITIONS: Tinnitus
Keywords: P50, Psychomotor Vigilance Test (PVT), Arousal, Reaction Time
MeSH Terms: conditions — Tinnitus | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- modafinil (Active Comparator)
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Modafinil — 200 mg/day, morning dose
  Arms: modafinil
Other: Placebo — Sugar pill once per day in the morning.
  Arms: Placebo

SUMMARY:
A study on the effects of the FDA approved drug Modafinil upon attention problems associated with tinnitus. This is considered to be a safe drug with few side effects. Each subject will be asked to participate in 3 sessions each lasting approximately 1 hour in which cognitive testing and recordings will be taken. The study involves each subject taking a 2- week supply of Modafinil and a 2- week supply of placebo. We hypothesize inattention related to thalamocortical dysrhythmia found in tinnitus can be reduced by Modafinil thus improving vigilance.

DETAILED DESCRIPTION:
Modafinil, a drug primarily used in the treatment for narcolepsy, is also being using in treating attention problems found in Attention Deficit Hyperactive Disorder (ADHD). This study will investigate the efficacy of Modafinil upon attention deficits found in tinnitus patients by assessing pre-attentional and attentional processes (e.g., the amplitude of auditory evoked responses and simple reaction time).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of tinnitus should be established by subject through exam and history performed by study physician in Ear, Nose and Throat (ENT) clinic.
* Subjects will be age 20 or older.
* Subjects should have tinnitus symptoms severe enough to seek medical attention.
* Subjects will have been seen in the Hearing and Balance Center at University of Arkansas for Medical Sciences (UAMS).
* Subjects will have had an audiogram.
* Signed informed consent.
* Women of childbearing potential must have a negative pregnancy test at screening and before being prescribed the study drug.
* Peripheral neuropathy.
* Hematologic (minimal values) at screening Absolute neutrophil count > 1,500 mm^3 Hemoglobin > 8.0 g/dl Platelet count > 100,000 mm^3

Exclusion Criteria:

Disease-Specific Concerns

* Subjects who have locally advanced breast cancer with skin ulceration will be excluded from this study due to the risk of worsening ulcers and healing difficulties
* Stage IV breast cancer
* Inflammatory breast cancer

General Medical Concerns

* Subjects with Echo Cardiogram performance status 2, 3, and 4 are not eligible for this study
* Allergy to any component of the treatment regimen
* Women who are breast feeding
* Pregnancy or refusal to use effective contraception while participating in this study
* Inability to comply with study and/or follow-up procedures
* Subjects with secondary malignancy other than superficial skin cancer (squamous cell carcinoma and basal cell carcinoma of the skin) should be excluded

Bevacizumab-Specific Concerns

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Blood pressure of > 150/100 mmHg. Essential hypertension well controlled with anti hypertensive is not an exclusion criterion
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix D)
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Presence of central nervous system or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating
* Urine protein: creatinine ratio >1.0 at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John L Dornhoffer, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from treatment clinic, seeking treatment for tinnitus.
Groups:
- Baseline, Modafinil 200 mg/Day, Placebo: Subjects are tested at baseline, then after Modafinil (200mg/day, a.m. administration) for 14 days, then after placebo (for 14 days).
- Baseline, Placebo, Modafinil 200 mg/Day: Subjects are tested after baseline, then after taking a sugar pill once per day in the morning for 14 days, and then after taking modafinil 200 mg/day for 14 days.
Period: Baseline (1 Day)
Arm/Group | Baseline, Modafinil 200 mg/Day, Placebo | Baseline, Placebo, Modafinil 200 mg/Day
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0
Period: Intervention 1 (14 Days)
Arm/Group | Baseline, Modafinil 200 mg/Day, Placebo | Baseline, Placebo, Modafinil 200 mg/Day
Started | 2 (One subject dropped out after baseline) | 3 (One subject dropped out after baseline)
Completed | 2 | 3
Not Completed | 0 | 0
Period: Intevention 2 (14 Days)
Arm/Group | Baseline, Modafinil 200 mg/Day, Placebo | Baseline, Placebo, Modafinil 200 mg/Day
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Subjects were tested at baseline, then entered either the modafinil or placebo condtion and then the remaining condition.
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The P50 Amplitude (i.e. Evoked Auditory Response Potential Recorded in Millivolts 50 Milliseconds After Sound Onset).
Description: P50 is an auditory evoked response potential sensitive to states of arousal.
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: milli volts
Groups:
- Baseline Testing.: Establish baseline levels of performance
- Modafinil: Subjects are tested after taking Modafinil (200mg/day, a.m. administration) for 14 days.
- Placebo: Subjects are tested after taking a sugar pill once per day in the morning for 14 days.
Arm/Group | Baseline Testing. | Modafinil | Placebo
Number analyzed (Participants) | 5 | 5 | 5
milli volts | 1.25 (.15) | 1.47 (.28) | 1.23 (.26)

2. Secondary Outcome: Simple Reaction Time (Attention)for Baseline, Modafinil and Placebo Arms.
Description: Simple reaction time to an auditory signal is a measure of attention.
Time Frame: 5 weeks
Measure: Mean (Standard Error); unit: milli seconds
Arm/Group | Baseline Testing. | Modafinil | Placebo
Number analyzed (Participants) | 5 | 5 | 5
milli seconds | 269.80 (12.64) | 268.12 (14.41) | 247.11 (8.14)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Baseline Testing. | Modafinil | Placebo
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of change in primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes